CLINICAL TRIAL: NCT01143948
Title: Insulin Therapy in the Inpatient Management of Cirrhotic Patients With Type 2 Diabetes
Brief Title: Various Insulin Regimens for Diabetic Inpatients With Cirrhosis Trial
Acronym: VIRDICT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Internal Medicine Department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC-T2D
Record Dates: First submitted 2010-06-10; First posted 2010-06-15 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-02

CONDITIONS: Type 2 Diabetes; Liver Cirrhosis
Keywords: Diabetes; Cirrhosis; Insulin; Inpatient
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Liver Cirrhosis; Diabetes Mellitus; Fibrosis; Insulin Resistance | interventions — Insulin Glargine; insulin glulisine; Insulin; insulin, pork; isophane insulin, pork drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 15 patient sliding scale regular insulin (Active Comparator)
  Interventions: Drug: Regular insulin
- 15 patient BBI NPH plus regular insulin (Active Comparator)
  Interventions: Drug: NPH & regular insulin
- 15 patients BBI Glargine plus Glulisine (Active Comparator)
  Interventions: Drug: Glargine & Glulisine

INTERVENTIONS:
Drug: Glargine & Glulisine — Basal Glargine & bolus Glulisine
  Other Names: lantus; apidra
  Arms: 15 patients BBI Glargine plus Glulisine
Drug: Regular insulin — Sliding scale regular insulin
  Other Names: actrapid
  Arms: 15 patient sliding scale regular insulin
Drug: NPH & regular insulin — Basal NPH & bolus regular insulin
  Other Names: mixtard
  Arms: 15 patient BBI NPH plus regular insulin

SUMMARY:
Liver disease is an important cause of death in type 2 diabetes. In the population-based Verona Diabetes Study cirrhosis was the fourth leading cause of death and accounted for 4.4% of diabetes-related deaths. In another prospective cohort study , cirrhosis accounted for 12.5% of deaths in patients with diabetes. In Egypt hepatitis C virus the commonest of cirrhosis here has a prevalence of 9.8% in the population with the greatest burden over national health care bills. Patients with cirrhosis & type 2 diabetes mellitus are always showing up in all hospital wards without a clear consensus of best management of their hyperglycemia.

DETAILED DESCRIPTION:
Best management of hyperglycemia in non-intensive care unit Cirrhotic patients with type 2 diabetes by different insulin regimens either sliding scale regular insulin or basal bolus insulin using NPH & regular insulin or Glargine & Glulisine.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized type 2 Diabetes Mellitus with liver cirrhosis
* Entry blood glucose (fasting or random) greater than 180 mg%

Exclusion Criteria:

* Type 1 Diabetes Mellitus
* Pregnancy
* Steroids: prednisone greater than 7.5mg/day or equivalent
* Serum Creatinine > 3 mg/dl
* Patients in intensive care units.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-04 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
optimal glycemic control in inpatient cirrhotics | 3-7 days

SECONDARY OUTCOMES:
Incidence of hypoglycemic episodes | 3-7 days

CONTACTS AND LOCATIONS:
Overall Officials: Ibtisam Z Eissa, MD, Study Chair — Cairo University; Mary N Rizk, MD, Study Director — Cairo Univerity; Ahmad A Khairy, MD, Study Director — Cairo University
Locations (1):
- Internal medicine hospital ,Cairo University, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Background] Balkau B, Eschwege E, Ducimetiere P, Richard JL, Warnet JM. The high risk of death by alcohol related diseases in subjects diagnosed as diabetic and impaired glucose tolerant: the Paris Prospective Study after 15 years of follow-up. J Clin Epidemiol. 1991;44(6):465-74. doi: 10.1016/0895-4356(91)90209-r. PMID 2037851
- [Background] de Marco R, Locatelli F, Zoppini G, Verlato G, Bonora E, Muggeo M. Cause-specific mortality in type 2 diabetes. The Verona Diabetes Study. Diabetes Care. 1999 May;22(5):756-61. doi: 10.2337/diacare.22.5.756. PMID 10332677
- [Result] Tolman KG, Fonseca V, Dalpiaz A, Tan MH. Spectrum of liver disease in type 2 diabetes and management of patients with diabetes and liver disease. Diabetes Care. 2007 Mar;30(3):734-43. doi: 10.2337/dc06-1539. No abstract available. PMID 17327353